CLINICAL TRIAL: NCT07035262
Title: Preoperative and Postoperative Changes in Serum Metabolome Dynamics in Colorectal Cancer Patients and Their Impact on Perioperative Clinical Outcomes
Brief Title: Impact of Pre- and Post-operative Serum Metabolome Dynamics in Colorectal Resection Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2025-364-01
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Colo-rectal Cancer
Keywords: colorectal cancer; postoperative complication; surgery; metabolites
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the colorectal cancer group: patients diagnosed with colorectal cancer
  Interventions: Other: serum metabolites

INTERVENTIONS:
Other: serum metabolites — serum metabolites before and after colorectal cancer surgery

SUMMARY:
The aim of this study is to systematically analyze the dynamic pattern of preoperative and postoperative serum metabolites in colorectal cancer patients through metabolomics technology, and to screen the key metabolites with statistical differences and explore their correlation with surgical interventions by combining the baseline characteristics of the patients with the perioperative clinical data; to further reveal the impact of surgery on the body's metabolic remodeling pattern, and to explore the potential biomarkers and regulatory pathways, providing a theoretical basis for elucidating the metabolic mechanism. Investigaters will further reveal the impact of surgery on metabolic remodeling, explore potential biomarkers and regulatory pathways, provide theoretical basis for elucidating the metabolic mechanism, and evaluate its clinical translational value (e.g., postoperative monitoring, targeted intervention, etc.), so as to lay the foundation for the subsequent basic research and precise treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Previous consent to participate;
* Blood drawn and serum samples extracted and preserved both preoperatively and postoperatively;
* Successful detection of metabolomics profiles from serum samples;
* Acceptance of a standard radical colorectal cancer procedure;
* Complete perioperative data available;
* Adults with a pathologic diagnosis of colorectal cancer

Exclusion Criteria:

* Have or have had a previous history of other malignancies;
* Have a history of radiotherapy treatment;
* Have a history of inflammatory bowel disease;
* Have a familial history of genetic disorders;
* Missing baseline data (age, BMI, gender, previous medical history, etc.);
* Failed to leave the hospital earlier than medically indicated;
* Failed to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | From the first day of surgery to two months after surgery
  Postoperative complications occurring within two months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Ethics committees require no data sharing due to patient privacy protection.